CLINICAL TRIAL: NCT02211859
Title: An Open Phase I Repeated Dose Escalation Study of BI 2536 BS Administered Intravenously in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: Dose Escalation Study of BI 2536 BS in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1216.2
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 2536

ARMS (1):
- BI 2536 (Experimental): single escalating dose, followed by repeated administration in patients with clinical benefit
  Interventions: Drug: BI 2536

INTERVENTIONS:
Drug: BI 2536

SUMMARY:
Primary: Maximum tolerated dose (MTD) Secondary: Determination of the pharmacokinetic profile of BI 2536. Assessment of safety and efficacy.

ELIGIBILITY:
Inclusion criteria:

* Patients with confirmed diagnosis of advanced, non resectable and/or metastatic solid tumours, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
* Evaluable tumour deposits
* Age 18 years or older
* Life expectancy of at least six months
* Written informed consent consistent with international conference of harmonization (ICH) - good clinical practice (GCP) and local legislation
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
* Full recovery from all therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies

Exclusion Criteria:

* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Pregnancy or breastfeeding
* Active infectious disease
* Known brain metastases
* Second malignancy requiring therapy
* Absolute neutrophil count less than 1500/mm3
* Platelet count less than 100 000/mm3
* Bilirubin greater than 1.5 mg/dl (> 26 μmol/L)
* Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg/dl (> 132 μmol/L)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) by occurrence of dose limiting toxicities (DLT) | up to 3 weeks

SECONDARY OUTCOMES:
Number of patients with drug-related adverse events | up to 24 days after last drug administration
  according to common terminology criteria for adverse events (CTCAE) 3.0
Number of patients with abnormal laboratory findings | up to 24 days after last drug administration
Change in Eastern Cooperative Oncology Group (ECOG) performance score | baseline, up to 24 days after last drug administration
Number of patients with clinically significant changes in vital signs | up to 24 days after last drug administration
Number of patients with objective tumor response | up to 24 days after last drug administration
Cmax (maximum concentration of the analyte in plasma) | up to 264 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 264 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 264 hours after drug administration
%AUC0-tz (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 264 hours after drug administration
λz (terminal rate constant in plasma) | up to 264 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 264 hours after drug administration
MRT (mean residence time of the analyte in the body after intravenous administration) | up to 264 hours after drug administration
CL (total clearance of the analyte in the plasma after intravascular administration) | up to 264 hours after drug administration
Vz (apparent volume of distribution during the terminal phase λz following an intravascular dose) | up to 264 hours after drug administration
Vss (apparent volume of distribution at steady state following intravascular administration) | up to 264 hours after drug administration

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing